CLINICAL TRIAL: NCT01869699
Title: Effects of Intravenous Acetaminophen on Body Temperature and Hemodynamic Responses in Febrile Critically Ill Adults: a Randomized Controlled Trial
Brief Title: Effects of Intravenous Acetaminophen on Body Temperature and Hemodynamic Responses in Febrile Critically Ill Adults
Acronym: ICUFeverAPAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCSF-ICUFever
Record Dates: First submitted 2013-05-31; First posted 2013-06-05 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-07

CONDITIONS: Fever; Critical Illness
Keywords: Fever; Acetaminophen; Critical Care; ICU; Febrile
MeSH Terms: conditions — Fever; Critical Illness | interventions — Acetaminophen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal saline placebo (Placebo Comparator): Normal saline 100 mLs intravenous, administered over 15 minutes
  Interventions: Drug: Placebo
- Acetaminophen (Experimental): Acetaminophen 1 gram/100 mLs intravenous, single dose administered over 15 minutes
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — acetaminophen 1 gram/100mLs intravenously administered over 15 minutes
  Other Names: Ofirmev
  Arms: Acetaminophen
Drug: Placebo — Normal saline placebo Normal saline 100 mLs intravenous, administered over 15 minutes
  Other Names: NS; 0.9% sodium chloride
  Arms: Normal saline placebo

SUMMARY:
The purpose of this study is to compare the effects of intravenous acetaminophen to placebo on body temperature and hemodynamic (heart rate and blood pressure) responses in febrile critically ill adult patients.

There are limited data to explain the variable and unpredictable antipyretic and hemodynamic response to acetaminophen in febrile ICU patients. The complex pathophysiology of critically ill patients, co-morbid conditions, the effect of multiple pharmacologic and non-pharmacologic care interventions, and/or the potential interferences with absorption of enteral or rectal formulations may be related to variations in the antipyretic response to acetaminophen. It is necessary for clinicians to have a better understanding of the therapy response and potential adverse effects of this commonly administered medication, especially the recently available IV formulation, in critically ill patients. Further research of the antipyretic response to acetaminophen in critically ill patients is warranted to inform evidence-based practice guidelines for fever management. Further randomized, placebo-controlled studies of hemodynamic responses to IV acetaminophen are also warranted.

Primary Hypothesis:

There is a significant reduction in time-weighted average core body temperature over 4 hours after administration of IV acetaminophen compared to placebo in febrile critically ill patients.

Secondary Hypotheses:

1. There is a significant reduction in time-weighted average heart rate over 4 hours after administration of IV acetaminophen compared to placebo in febrile critically ill patients.
2. There is a significant reduction in time-weighted mean arterial pressure over 4 hours after administration of IV acetaminophen compared to placebo in febrile critically ill patients.

Adult patients with fever (≥ 38.3ºCentigrade/101ºFarenheit) in the intensive care unit will be screened for eligibility and enrolled after informed consent. Patients will be randomized to receive IV acetaminophen 1 gram or normal saline 100 mLs. Body temperature, heart rate, and blood pressure will be measured at baseline and during the 4 hours post study drug administration.

DETAILED DESCRIPTION:
Adult patients with fever (≥ 38.3ºCentigrade (C)/101ºFarenheit(F)) in the intensive care unit will be screened for eligibility and approached for informed consent. Enrolled patients will be stratified based on the leading etiology of their fever: either neurologic injury or infection and then randomized to receive IV acetaminophen 1 gram or normal saline 100 milliliters (mLs). Core body temperature will be measured using a zero-heat flow thermometry system (non-invasive, small disk on forehead). Patients will be monitored and data collected during the 4-hour post study drug administration period. A rescue protocol will be implemented if the temperature reaches ≥ 40 ºC during the study period and includes notification of primary team provider by the nurse and the pharmacist will contact them to inform the provider of study group (acetaminophen or placebo). The provider can decide whether to order antipyretic medication or physical cooling interventions at that time.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Patient in an intensive care unit
* Weight greater or equal to 50 kgs
* Fever: core body temperature greater than or equal to 38.3 degrees Celsius
* Clinically stable: no active resuscitation with fluids, blood products, or dose increases of vasoactive medications within 1 hour of study drug administration

Exclusion Criteria:

* Acetaminophen hypersensitivity
* Acute liver failure or acute liver injury
* Heat stroke, malignant hyperthermia, neuroleptic malignant syndrome
* Therapeutic cooling, physical cooling, extracorporeal blood circuit therapies
* Administration of acetaminophen-containing medications, non-steroidal anti-inflammatory drugs, or aspirin greater than 81 mg within specified times per drug prior to fever presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A. Puntillo, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Medical Center, San Francisco, California
  - University of California, San Francisco Medical Center, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laupland KB, Zahar JR, Adrie C, Schwebel C, Goldgran-Toledano D, Azoulay E, Garrouste-Orgeas M, Cohen Y, Jamali S, Souweine B, Darmon M, Timsit JF. Determinants of temperature abnormalities and influence on outcome of critical illness. Crit Care Med. 2012 Jan;40(1):145-51. doi: 10.1097/CCM.0b013e31822f061d. PMID 21926588
- [Background] Lee BH, Inui D, Suh GY, Kim JY, Kwon JY, Park J, Tada K, Tanaka K, Ietsugu K, Uehara K, Dote K, Tajimi K, Morita K, Matsuo K, Hoshino K, Hosokawa K, Lee KH, Lee KM, Takatori M, Nishimura M, Sanui M, Ito M, Egi M, Honda N, Okayama N, Shime N, Tsuruta R, Nogami S, Yoon SH, Fujitani S, Koh SO, Takeda S, Saito S, Hong SJ, Yamamoto T, Yokoyama T, Yamaguchi T, Nishiyama T, Igarashi T, Kakihana Y, Koh Y; Fever and Antipyretic in Critically ill patients Evaluation (FACE) Study Group. Association of body temperature and antipyretic treatments with mortality of critically ill patients with and without sepsis: multi-centered prospective observational study. Crit Care. 2012 Feb 28;16(1):R33. doi: 10.1186/cc11211. PMID 22373120
- [Background] Laupland KB, Shahpori R, Kirkpatrick AW, Ross T, Gregson DB, Stelfox HT. Occurrence and outcome of fever in critically ill adults. Crit Care Med. 2008 May;36(5):1531-5. doi: 10.1097/CCM.0b013e318170efd3. PMID 18434882
- [Background] Circiumaru B, Baldock G, Cohen J. A prospective study of fever in the intensive care unit. Intensive Care Med. 1999 Jul;25(7):668-73. doi: 10.1007/s001340050928. PMID 10470569
- [Background] Frankenfield DC, Smith JS Jr, Cooney RN, Blosser SA, Sarson GY. Relative association of fever and injury with hypermetabolism in critically ill patients. Injury. 1997 Nov-Dec;28(9-10):617-21. doi: 10.1016/s0020-1383(97)00117-4. PMID 9624339
- [Background] Thompson HJ, Kagan SH. Clinical management of fever by nurses: doing what works. J Adv Nurs. 2011 Feb;67(2):359-70. doi: 10.1111/j.1365-2648.2010.05506.x. Epub 2010 Nov 2. PMID 21044137
- [Background] Niven DJ, Stelfox HT, Laupland KB. Antipyretic therapy in febrile critically ill adults: A systematic review and meta-analysis. J Crit Care. 2013 Jun;28(3):303-10. doi: 10.1016/j.jcrc.2012.09.009. Epub 2012 Nov 14. PMID 23159136
- [Background] de Maat MM, Tijssen TA, Bruggemann RJ, Ponssen HH. Paracetamol for intravenous use in medium--and intensive care patients: pharmacokinetics and tolerance. Eur J Clin Pharmacol. 2010 Jul;66(7):713-9. doi: 10.1007/s00228-010-0806-5. Epub 2010 Mar 19. PMID 20300741
- [Background] Kett DH, Breitmeyer JB, Ang R, Royal MA. A randomized study of the efficacy and safety of intravenous acetaminophen vs. intravenous placebo for the treatment of fever. Clin Pharmacol Ther. 2011 Jul;90(1):32-9. doi: 10.1038/clpt.2011.98. Epub 2011 May 4. PMID 21544074
- [Background] Mackenzie I, Forrest K, Thompson F, Marsh R. Effects of acetaminophen administration to patients in intensive care. Intensive Care Med. 2000 Sep;26(9):1408. doi: 10.1007/s001340000614. No abstract available. PMID 11089781
- [Background] Boyle M, Hundy S, Torda TA. Paracetamol administration is associated with hypotension in the critically ill. Aust Crit Care. 1997 Dec;10(4):120-2. doi: 10.1016/s1036-7314(97)70414-4. PMID 9708071
- [Background] Boyle M, Nicholson L, O'Brien M, Flynn GM, Collins DW, Walsh WR, Bihari D. Paracetamol induced skin blood flow and blood pressure changes in febrile intensive care patients: An observational study. Aust Crit Care. 2010 Nov;23(4):208-14. doi: 10.1016/j.aucc.2010.06.004. Epub 2010 Jul 22. PMID 20655241
- [Background] Hersch M, Raveh D, Izbicki G. Effect of intravenous propacetamol on blood pressure in febrile critically ill patients. Pharmacotherapy. 2008 Oct;28(10):1205-10. doi: 10.1592/phco.28.10.1205. PMID 18823215

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Saline Placebo | Acetaminophen
Started | 21 | 20
Completed | 20 | 20
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline Placebo | Acetaminophen | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (13) | 58 (15) | 57.5 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 17 | 14 | 31
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared] — Body Mass Index (BMI) units of measure are kilograms per meter squared
  kilograms per meter squared | 31 (7) | 29 (5) | 30 (6)
Primary ICU diagnosis [Count of Participants; unit: Participants]
  Number of patients with Medical diagnoses | 6 | 6 | 12
  Number of patients with Surgical diagnoses | 4 | 2 | 6
  Number of patients iwth Neurologic diagnoses | 10 | 12 | 22
Acute Physiologic and Chronic Health Evaluation (APACHE) II score [Mean (Standard Deviation); unit: scores on a scale] — Acute Physiologic and Chronic Health Evaluation (APACHE) II is a severity-of-disease classification system (Knaus et al., 1985), one of several ICU scoring systems. It is applied within 24 hours of admission of a patient to an intensive care unit (ICU): an integer score from 0 to 71 is computed based on several measurements; higher scores correspond to more severe disease.
  scores on a scale | 24 (6) | 24 (6) | 24 (6)
Number of patients with infectious and noninfectious etiology of fever [Count of Participants; unit: Participants]
  Number of patients with Infectious etiology | 15 | 15 | 30
  Number of patients with Noninfectious etiology | 5 | 5 | 10
Number of patients receiving types of medication infusions [Count of Participants; unit: Participants]
  Number of patients on vasopressor infusions | 6 | 4 | 10
  Number of patients on vasodilator infusions | 2 | 2 | 4
  Number of patients on sedative infusions | 9 | 8 | 17
  Number of patients on analgesic infusions | 3 | 1 | 4
  Number of patients on no medication infusions | 0 | 5 | 5
Number of patients with sepsis [Count of Participants; unit: Participants] — Sepsis was defined as new confirmed or suspected infection and 2 or more systemic inflammatory response syndrome (SIRS) criteria. (Dellinger RP, Levy MM, et al. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Medicine 2013; 39: 165-228.)
  Participants | 14 | 13 | 27
Number of patients receiving Mechanical Ventilation [Count of Participants; unit: Participants] | 15 | 12 | 27
Mode of ventilation [Count of Participants; unit: Participants]
  Number of patients on Pressure Support | 11 | 10 | 21
  Number of patients on Assist Control | 4 | 2 | 6
  Number of patients NOT on mechanical ventilation | 5 | 8 | 13
Temperature of room [Mean (Standard Deviation); unit: degrees Celsius] | 21.5 (1.4) | 21.4 (1.2) | 21.4 (1.3)
Core body temperature [Mean (Standard Deviation); unit: degrees Celsius] | 38.6 (0.5) | 38.4 (0.3) | 38.5 (0.4)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] | 93 (15) | 90 (14) | 91.5 (14.5)
systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 135 (26) | 151 (26) | 143 (26)
diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 64 (13) | 73 (15) | 67.5 (14)
mean arterial pressure [Mean (Standard Deviation); unit: mm Hg] | 89 (16) | 100 (20) | 94.5 (18)
respiratory rate [Mean (Standard Deviation); unit: breaths per minute] | 24 (5) | 20 (6) | 22 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Core Body Temperature
Description: time-weighted average core body temperature over 4 hours. Core temperature was measured every 5 minutes times 4, and then every 15 minutes over the following 4 hours from the time of study drug administration. The sum of the core temperature values was divided by time in minutes.
Time Frame: Baseline to 4 hours post study drug administration
Population: Patients in an ICU with fever, weighed > 50kg and did not meet any exclusion criteria.
Measure: Mean (Standard Error); unit: degrees Celsius
Arm/Group | Normal Saline Placebo | Acetaminophen
Number analyzed (Participants) | 20 | 20
degrees Celsius | 38.4 (0.1) | 37.9 (0.1)
Statistical Analysis 1: Comparison: Normal Saline Placebo vs Acetaminophen; We estimated that 20 patients per group would provide 80% power for detecting a difference in means of 0.6 degrees Celsius, with a pooled SD of 0.67 degrees, using a two group t test and a two sided alpha level of 0.05. A previous RCT of IV acetaminophen in healthy male volunteers with induced fever found a core temperature difference of 0.60 degrees with a common SD of 0.67 degrees Celsius; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.76 to -0.18]

2. Secondary Outcome: Heart Rate
Description: time-weighted average heart rate over 4 hours. Heart rate was measured every 5 minutes times 4, and then every 15 minutes over the following 4 hours from the time of study drug administration. The sum of the heart rate values was divided by time in minutes.
Time Frame: Baseline to 4 hours post study drug administration
Population: Patients in the ICU with fever, weight of > 50kg and no exclusion criteria met.
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Normal Saline Placebo | Acetaminophen
Number analyzed (Participants) | 20 | 20
beats per minute | 92 (2) | 87 (2)
Statistical Analysis 1: Comparison: Normal Saline Placebo vs Acetaminophen; Test type: Superiority; p = 0.03, ANCOVA; Mean Difference (Final Values) = -6, 95% CI 2-sided [-10 to -1]

3. Secondary Outcome: Systolic Blood Pressure
Description: time-weighted average systolic blood pressure over 4 hours. Systolic blood pressure was measured every 5 minutes times 4, and then every 15 minutes over the following 4 hours from the time of study drug administration. The sum of the systolic blood pressure values was divided by time in minutes.
Time Frame: Baseline to 4 hours post study drug administration
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Normal Saline Placebo | Acetaminophen
Number analyzed (Participants) | 20 | 20
mm Hg | 143 (3) | 127 (3)
Statistical Analysis 1: Comparison: Normal Saline Placebo vs Acetaminophen; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Final Values) = -17, 95% CI 2-sided [-25 to -8]

4. Secondary Outcome: Respiratory Rate
Description: time weighted average for respiratory rate over 4 hours. Respiratory rate was measured every 5 minutes times 4, and then every 15 minutes over the following 4 hours from the time of study drug administration. The sum of the respiratory rate values was divided by time in minutes.
Time Frame: Baseline to 4 hours post study drug administration
Population: Patients in the ICU with fever, weight of > 50kg and no exclusion criteria met.
Measure: Mean (Standard Error); unit: breaths per minute
Arm/Group | Normal Saline Placebo | Acetaminophen
Number analyzed (Participants) | 20 | 20
breaths per minute | 22 (1) | 21 (1)
Statistical Analysis 1: Comparison: Normal Saline Placebo vs Acetaminophen; Test type: Superiority; p = 0.42, ANCOVA; Mean Difference (Final Values) = -1, 95% CI 2-sided [-4 to 12]

5. Secondary Outcome: 2-hour Change Over Time Core Temperature
Description: change over time core temperature after study drug administration (adjusted to baseline core temperature)
Time Frame: 2 hours
Measure: Mean (Standard Error); unit: degrees Celsius
Arm/Group | Normal Saline Placebo | Acetaminophen
Number analyzed (Participants) | 20 | 20
degrees Celsius | -0.01 (1.3) | -0.8 (1.3)
Statistical Analysis 1: Comparison: Normal Saline Placebo vs Acetaminophen; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1 to -0.3]

6. Secondary Outcome: 2-hour Change Over Time Systolic Blood Pressure
Description: 2-hour change over time SBP from study drug administration (means adjusted to baseline SBP)
Time Frame: Baseline to 2 hours
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Normal Saline Placebo | Acetaminophen
Number analyzed (Participants) | 20 | 20
mm Hg | -0.1 (5) | -24 (5)
Statistical Analysis 1: Comparison: Normal Saline Placebo vs Acetaminophen; Test type: Superiority; p = 0.001, ANCOVA; Mean Difference (Final Values) = -24, 95% CI 2-sided [-38 to -10]

7. Secondary Outcome: 2-hour Change Over Time Heart Rate
Description: 2-hour change over time heart rate from time of study drug administration (means adjusted to baseline HR)
Time Frame: Baseline to 2 hours
Measure: Mean (Standard Error); unit: BPM
Arm/Group | Normal Saline Placebo | Acetaminophen
Number analyzed (Participants) | 20 | 20
BPM | 2 (2) | -6 (2)
Statistical Analysis 1: Comparison: Normal Saline Placebo vs Acetaminophen; Test type: Superiority; p = 0.02, ANCOVA; Mean Difference (Final Values) = -8, 95% CI 2-sided [-15 to -1]

ADVERSE EVENTS:
Arm/Group | Normal Saline Placebo | Acetaminophen
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
The generalizability of our findings is limited due to the use of a single site and our sample size was modest. Also, patients in this study had baseline stable and normal or high BP, so unclear if same results in patients with unstable or low BP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No